CLINICAL TRIAL: NCT03755544
Title: Salmeterol/Fluticasone Easyhaler in the Treatment of Asthma and COPD; a Non-interventional Switch Study to Evaluate the Impact on Clinical Effects, Patient's Satisfaction, Preference and Use of Easyhaler
Brief Title: Salmeterol/Fluticasone Easyhaler in the Treatment of Asthma and COPD
Acronym: SUNNY
Status: Completed | Type: Observational
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 3106013
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma patients: Male or female patients with diagnosed asthma who have been using salmeterol/fluticasone propionate combination treatment for at least 3 months before the beginning of the study, and for whom the decision has already been made to switch to Salmeterol/fluticasone Easyhaler.
  During the study, the Salmeterol/fluticasone Easyhaler will be used according to the local Summary of Product Characteristics (SmPC).
- COPD patients: Male or female patients with diagnosed COPD who have been using salmeterol/fluticasone propionate combination treatment for at least 3 months before the beginning of the study, and for whom the decision has already been made to switch to Salmeterol/fluticasone Easyhaler.
  During the study, the Salmeterol/fluticasone Easyhaler will be used according to the local Summary of Product Characteristics (SmPC).

SUMMARY:
A non-interventional study to assess the clinical effectiveness of Salmeterol/fluticasone Easyhaler to achieve and maintain asthma or COPD control.

DETAILED DESCRIPTION:
A prospective, open-label, non-interventional, multicentre study in adult patients with asthma or COPD who are treated with Salmeterol/fluticasone Easyhaler. During the study the Salmeterol/fluticasone Easyhaler will be used according to the Summary of Product Characteristics. Clinical effectiveness of the treatment will be evaluated with change in asthma or COPD symptoms during 12 weeks treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female patients with asthma or COPD who have been using salmeterol/fluticasone propionate combination treatment for at least 3 months before the study
2. Age ≥18 years.
3. Written informed consent obtained.

Main Exclusion Criteria:

1. Pregnant or lactating female patients.
2. Participation in other clinical studies during the study.
3. Known hypersensitivity (allergy) to salmeterol, fluticasone propionate or the excipient lactose
4. Any significant medical disease or condition or other factor that might interfere with study assessments or study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients will be enrolled by physicians from outpatient clinics
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 12 weeks
  A multiple-choice questionnaire for patients with asthma, each choice is assigned a score 1-5. There are 5 questions to answer. The total score is calculated, ranging between 5 and 25. Lower scores indicate worse asthma control.
COPD Assessment Test (CAT) | 12 weeks
  A bipolar questionnaire for patients with COPD, there are 8 questions with 2 answers showing different extremes, respondents choose the numbered answer that reflects their opinion (in the range 0-5). The total score is calculated and ranges between 0 and 40. Higher scores indicate worse COPD control.

SECONDARY OUTCOMES:
Asthma symptom control assessment | 12 weeks
  A dichotomous questionnaire for patients with asthma, there are 4 questions with 'Yes' or 'No' answers, respondents choose the answer that reflects their opinion. A great number of 'Yes' answers indicate worse asthma control.
Forced expiratory volume in one second (FEV1) | 12 weeks
  from spirometry
Feeling of Satisfaction with Inhaler questionnaire (FSI-10) | 12 weeks
  patient's satisfaction with inhaler
A questionnaire to assess Physician's/nurse's perception of Salmeterol/fluticasone Easyhaler overall use | 12 weeks
  A multiple-choice questionnaire for the physician/nurse, completed for each patient. Evaluation will be by frequency tables and summary statistics.
Mini-AQLQ questionnaire | 12 weeks
  A multiple-choice questionnaire for patients with asthma, each choice is assigned a score 1-7. There are 15 questions to answer. The total score is calculated and ranges between 15 and 105. Lower scores indicate worse quality of life.
Health care utilisation questionnaire | 24 weeks
  A dichotomous questionnaire for all patients, there are 6 questions, with 'Yes' or 'No' answers, to collect health care use. Evaluation will be by frequency tables and summary statistics.
Modified Medical Research Council (mMRC) dyspnea questionnaire | 12 weeks
  A bipolar questionnaire for patients with COPD, there is one question with 5 choices between two extremes, respondents choose the answer that reflects their opinion (in the range 0-4).. Higher scores indicate worse dyspnea symptoms.
Symptom burden and exacerbation risk assessment (ABCD classification) | 12 weeks
  Patients will be assessed by the physician, based on symptoms and exacerbation history according to the ABCD classification scheme (GOLD, 2018).
Forced vital capacity (FVC) | 12 weeks
  from spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Orion Pharma Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Lungenpraxis, Hamburg, Germany